CLINICAL TRIAL: NCT01442246
Title: Phase III Randomised Trial to Evaluate the Benefit of Adjuvant Hormonal Treatment With Leuprorelin Acetate (Eligard® 45 mg) for 24 Months After Radical Prostatectomy in Patients With High Risk of Recurrence.
Brief Title: Evaluation of Adjuvant Hormonal Treatment for 24 Months After Radical Prostatectomy in High Risk of Recurrence Patients.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFU-GETUG 20 - UC-0160/1003; 2010-022037-29 (EudraCT Number)
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastases
Keywords: Benefit of; adjuvant; treatment; prostatectomy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant treatment (Experimental): Leuproreline acetate
  Interventions: Drug: Leuprorelin Acetate
- Surveillance (No Intervention): Surveillance

INTERVENTIONS:
Drug: Leuprorelin Acetate — Leuprorelin Acetate 45 mg, one injection every 6 months for 24 months
  Other Names: Eligard®
  Arms: Adjuvant treatment

SUMMARY:
PRINCIPAL OBJECTIVE: Evaluation of effectiveness in terms of survival without metastases to 10 years, of adjuvant hormonal treatment with leuprorelin acetate (Eligard® 45 mg) for 24 months after radical prostatectomy in patients with high risk of recurrence.

SECONDARY OBJECTIVE(S):

* PSA evolution
* Evaluation of testosterone level
* Specific survival
* Overall survival
* Tolerance
* Quality of life (QLQ-C30 questionnaires)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have received the information leaflet and signed the consent form
2. ≥18 years of age with a life expectancy of at least 10 years
3. Performance Status (ECOG) ≤2
4. Radical prostatectomy (RP) with or without extended pelvic lymphadenectomy in the 3 months preceding inclusion
5. Histologically confirmed prostatic adenocarcinoma
6. Patients R0, N0 or Nx or N+ (≤ 2 nodes among nodes removed), M0 and with at least one of the following criteria:

   * postoperative Gleason score >7
   * postoperative Gleason score =7 with the presence of high-grade Gleason patterns
   * pT3b patients
7. Postoperative PSA <0.1 ng/mL (dosage perform within 2 months after surgery)
8. Neutrophils ≥1500/mm³, platelets ≥100000/mm³
9. Bilirubin ≤ upper normal limit (this will not apply to subjects with Gilbert's syndrome, persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology); ASAT and ALAT ≤1.5 times upper normal limit; Creatinine <140 µmol/l (or clearance >60 mL/min)
10. Patients affiliated to a social security scheme

Exclusion Criteria:

1. Previous treatments for prostatic adenocarcinoma (HT or orchiectomy or CT)
2. Presence of metastases:

   * positive bone scintigraphy, including Patients with medullary compression and/or
   * abdominal-pelvic CT scan or MRI showing lymph node and/or visceral involvement
3. History of cancer, with the exception of basal cell carcinoma or any other cancer treated in the 5 years before inclusion and in complete remission
4. Incompatible concomitant treatment(s)
5. Hypersensitivity to other GnRH agonists and/or any of the excipients of Eligard®
6. Any illness or problem including geographic, psychiatric or psychological which is incompatible with being monitored during the trial
7. Persons deprived of their freedom or under supervision (including guardianship),
8. Patients already included in another therapeutic trial with an experimental drug or having been given an experimental drug within a period of 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The principal criterion is the evaluation of effectiveness in terms of survival without metastases to 10 years, of adjuvant treatment with leuprorelin acetate (Eligard® 45 mg) for 24 months after radical prostatectomy. | The principal criterion will be evaluated 12 years after the inclusion of the first patient.

CONTACTS AND LOCATIONS:
Overall Officials: François ROZET, MD, Study Director — Montsouris Institute, Paris; Stephane Culine, Prof, MD, Study Chair — Saint-Louis Hospital, Paris, France
Locations (35):
- France (35):
  - Clinique Victor Pauchet, Amiens
  - Chu Besancon, Besançon
  - Chu Bordeaux- Hopital Pellegrin, Bordeaux
  - Institut Bergonie, Bordeaux
  - Chru de Brest, Brest
  - Hopital Henri Mondor, Créteil
  - Chu Bocage, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Chru Lille, Lille
  - Chu Limoges, Limoges
  - Hopital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Nord, Marseille
  - Clinique Beausoleil, Montpellier
  - Hopital Lapeyronie, Montpellier
  - Chu de Nancy, Nancy
  - Chu Nantes, Nantes
  - Chu Pasteur, Nice
  - Chu Caremeau, Nîmes
  - Hopital Saint Louis, Paris
  - Hopital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - HEGP, Paris
  - Hopital Tenon, Paris
  - Hopital Pitie Salpetriere, Paris
  - Chu La Miletrie, Poitiers
  - Institut Jean Godinot, Reims
  - Chu Pontchaillou, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Hopsitalier Prive - Polyclinique Du Littoral, Saint-Brieuc
  - Clinique Mutualiste, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Hopitaux Civils de Colmar, Strasbourg
  - Hopital Foch, Suresnes
  - Chu Rangueil, Toulouse